CLINICAL TRIAL: NCT01507272
Title: A Randomised, Double-blind, Placebo-controlled, Dose Escalation Trial of Single Doses of NNC90-1170 to Assess Tolerability, Pharmacokinetics, Pharmacodynamics and Absolute Bioavailability in Healthy Male Subjects
Brief Title: Safety and Tolerability of Liraglutide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1149
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (liraglutide) (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Administered as 5 single s.c. (under the skin) doses - 1.25, 2.5, 5, 10 and 20 mcg/kg once daily - in ascending order
  Other Names: NNC 90-1170
  Arms: NNC 90-1170 (liraglutide)
Drug: liraglutide — Subjects receiving the dose level 5 mcg/kg s.c. will in addition receive, after a wash-out of at least 7 days, a single i.v. (into the vein) dose of 5 mcg/kg
  Other Names: NNC 90-1170
  Arms: NNC 90-1170 (liraglutide)
Drug: placebo — Administered s.c. After a wash-out of at least 7 days, a single i.v. (into the vein) dose is administered
  Arms: Placebo
Drug: placebo — Administered as 5 single s.c. (under the skin) doses - 1.25, 2.5, 5, 10 and 20 mcg/kg once daily - in ascending order
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess the safety and tolerability (maximum tolerated dose) after five ascending single doses of NNC 90-1170 (liraglutide).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects of any ethnic origin
* Written informed consent obtained. (The subject must give signed informed consent before any trial-related activities. Trial-related activities are any procedures that would not have been performed during the normal management of the subject)
* Good general health based on medical history, physical and laboratory examinations, incl. ECG (electrocardiogram)
* Body mass index within the range 20-27 kg/m^2, inclusive

Exclusion Criteria:

* Any clinically significant abnormal laboratory test results or clinically significant abnormal ECG
* History of alcoholism or drug addiction; positive results in the plasma urine screens for illicit drug
* Alcohol intake within 48 hours of visit
* Hepatitis B surface antigen (HBsAg), Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies
* History of significant drug allergy or drug hypersensitivity
* Smoke 5 cigarettes or more, or the equivalent per day and is unable to refrain from smoking during the 3 days prior to the dosing day and during the confinement period
* Subjects who drink more than 8 cups of tea/coffee per day

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 1999-03; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve)

SECONDARY OUTCOMES:
Cmax, maximum concentration
tmax, time to maximum concentration
t½, terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manchester, United Kingdom

REFERENCES:
- [Result] Elbrond B, Jakobsen G, Larsen S, Agerso H, Jensen LB, Rolan P, Sturis J, Hatorp V, Zdravkovic M. Pharmacokinetics, pharmacodynamics, safety, and tolerability of a single-dose of NN2211, a long-acting glucagon-like peptide 1 derivative, in healthy male subjects. Diabetes Care. 2002 Aug;25(8):1398-404. doi: 10.2337/diacare.25.8.1398. PMID 12145241
- [Result] Agerso H, Vicini P. Pharmacodynamics of NN2211, a novel long acting GLP-1 derivative. Eur J Pharm Sci. 2003 Jun;19(2-3):141-50. doi: 10.1016/s0928-0987(03)00073-3. PMID 12791417
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com